CLINICAL TRIAL: NCT00984126
Title: Safety and Efficacy of N8 in Prevention and On-demand Treatment of Bleeding Episodes in Subjects With Haemophilia A
Brief Title: Safety and Efficacy of Turoctocog Alfa (N8) in Prevention and On-demand Treatment of Bleeding Episodes in Subjects With Haemophilia A: An Extension to Trials NN7008-3543, NN7008-3545, NN7008-3600, NN7008-3893 and NN7008-4015
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3568; 2008-005945-46 (EudraCT Number); U1111-1111-9377 (Other: WHO); JapicCTI-101357 (Registry Identifier: JAPIC)
Record Dates: First submitted 2009-09-21; First posted 2009-09-25 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Turoctocog alfa (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — The preventative treatment is administered intravenously (i.v.) at specific intervals either every second day or three times a week. Bleeding treatment will be administered if a bleed should occur.
Drug: turoctocog alfa — Treatment is administered intravenously (i.v.) during bleeds and occasionally as a preventative treatment (e.g. before physical activity)

SUMMARY:
This trial is conducted in Asia, Europe, Japan, Oceania, North America and South America.

The aim of the trial is to investigate the safety and efficacy of turoctocog alfa (N8) in Haemophilia A patients.

The trial is an extension to trials NN7008-3543 (start: March 2009, stop: September 2011) and NN7008-3545 (start: May 2010, stop: November 2011) and the pharmacokinetic trials NN7008-3600 (start: November 2010, stop: October 2011), NN7008-3893 (start: June 2011, stop: September 2011) and NN7008-4015 (start: August 2012, stop: March 2013).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent obtained before any trial-related activities
* Completion of trial NN7008-3543 or paediatric trial NN7008-3545 or Japanese trial NN7008-3600 or pharmacokinetic trial NN7008-3893 or NN7008-4015

Exclusion Criteria:

* Previous participation in the current trial (defined as withdrawal) or withdrawn subjects from NN7008-3522, NN7008-3543, NN7008-3545, NN7008-3600, NN7008-3893 or NN7008-4015 after administration of trial product

Ages: 6 Months to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-10-26 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (55):
- United States (13):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Spokane, Washington
- Brazil (4):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Rio de Janeiro
- Croatia (2):
  - Novo Nordisk Investigational Site, Split
  - Novo Nordisk Investigational Site, Zagreb
- Germany (4):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hanover
- Israel (2):
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (5):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
- Novo Nordisk Investigational Site, Riga, Latvia
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Poland (2):
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, İzmit
  - Novo Nordisk Investigational Site, Samsun
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester

REFERENCES:
- [Result] Ozelo M, Misgav M, Abdul-Karim F, Lentz S, Martin-Salces M, Matytsina I, Saugstrup T, Santagostino E. Stabilization of turoctocog alfa dose administered in a preventive regimen: 3-year interim results of the guardianTM-2 extension trial. Haemophilia - Special Issue: Abstracts of the WFH 2014 World Congress, May 11-15, Melbourne, Australia; 20 (3): 1-200
- [Result] Recht M, Lentz S, Zupancic-Salek S, Matytsina I, Landorph A, Saugstrup T. Factor VIII Dosing and Preventive Efficacy in Obese Patients with Hemophilia (BMI =30 kg/m2) - a Post-Hoc Sub-Analysis of the guardian™ Trials. American Society of Hematology - 56th Annual Meeting (ASH); Country: US City: San Francisco, CA
- [Result] Ozelo M, Misgav M, Abdul Karim F, Lentz SR, Martin-Salces M, Matytsina I, Saugstrup T, Santagostino E. Long-term patterns of safety and efficacy of bleeding prophylaxis with turoctocog alfa (NovoEight((R)) ) in previously treated patients with severe haemophilia A: interim results of the guardian() 2 extension trial. Haemophilia. 2015 Sep;21(5):e436-9. doi: 10.1111/hae.12737. Epub 2015 Jun 8. No abstract available. PMID 26058730
- [Result] Lentz SR, Cerqueira M, Janic D, Kempton C, Matytsina I, Misgav M, Oldenburg J, Ozelo M, Recht M, Rosholm A, Savic A, Suzuki T, Tiede A, Santagostino E. Interim results from a large multinational extension trial (guardian() 2) using turoctocog alfa for prophylaxis and treatment of bleeding in patients with severe haemophilia A. Haemophilia. 2016 Sep;22(5):e445-9. doi: 10.1111/hae.12990. Epub 2016 Jun 13. No abstract available. PMID 27291066
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were enrolled at 52 sites in 19 countries:Brazil (4 sites), Croatia (2), Germany (3), Israel (1), Italy (2), Japan (5), Latvia (1), Lithuania (1), Macedonia (1), Malaysia (1), Poland (2), Russian Federation (2), Serbia (5), Spain (2), Switzerland (1), Taiwan (1), Turkey (5), the United Kingdom (1) and the United States (12).
Pre-assignment Details: Subjects completing 1 of the trials NN7008-3543 (NCT00840086),NN7008-3545 (NCT01138501),NN7008-3600 (NCT01238367),NN7008-3893 (NCT01365520) and NN7008-4015 (NCT01692925) could continue treatment with turoctocog alfa in the extension trial (NN7008-3568). Both new subjects and those from main trial (NN7008-3568) could enter the on-demand sub-trial.
Groups:
- Small Children (0 - <6 Years): Subjects (0-<6 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during the trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day,20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in the relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in the relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016)
- Older Children (6 - <12 Years): Subjects (6-<12 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
- Adolescents (12 - <18 Years): Subjects (12-<18 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly.On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
- Adults (≥18 Years): Subjects (≥18 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day,20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
Period: Overall Study
Arm/Group | Small Children (0 - <6 Years) | Older Children (6 - <12 Years) | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Started | 27 | 28 | 23 | 135
Completed | 20 | 20 | 16 | 76
Not Completed | 7 | 8 | 7 | 59
Not completed — Protocol Violation | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Choose to join Pathfinder trial™ + other | 7 | 7 | 3 | 46
Not completed — Withdrawal criteria | 0 | 1 | 3 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set includes all dosed patients with data after dosing.
Groups:
- Adolescents (12 - <18 Years): Subjects (12-<18 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
- Total: Total of all reporting groups
Arm/Group | Small Children (0 - <6 Years) | Older Children (6 - <12 Years) | Adolescents (12 - <18 Years) | Adults (≥18 Years) | Total
Number analyzed (Participants) | 27 | 28 | 23 | 135 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (1.4) | 9.0 (1.8) | 14.9 (1.7) | 32.0 (11.5) | 23.6 (14.6)
Age, Customized [Number; unit: participants]
  Small children (0 - <6 years) | 27 | 0 | 0 | 0 | 27
  Older children (6 - <12 Years) | 0 | 28 | 0 | 0 | 28
  Adolescents (12 - <18 Years) | 0 | 0 | 23 | 0 | 23
  Adults (≥18 Years) | 0 | 0 | 0 | 135 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 27 | 28 | 23 | 135 | 213

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Development of FVIII Inhibitors (Greater Than or Equal to 0.6 Bethesda Units (BU)/mL)
Description: The frequency of inhibitors was calculated as number of patients with inhibitors during the trial divided by number of patients in the trial. This endpoint was measured during the trial.
Time Frame: After 90 months
Population: Full analysis set
Measure: Number; unit: subjects
Arm/Group | Small Children (0 - <6 Years) | Older Children (6 - <12 Years) | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 27 | 28 | 23 | 135
subjects | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Small Children (0 - <6 Years) vs Older Children (6 - <12 Years) vs Adolescents (12 - <18 Years) vs Adults (≥18 Years); A one-sided 95% upper confidence limit was based on an exact calculation for a binomial distribution; Test type: Superiority or Other; Incidence rate = 0, 95% CI 1-sided [upper limit 1.4]

2. Secondary Outcome: Frequency of Adverse Events and Serious Adverse Events
Description: The number of adverse events and serious adverse events reported during the main trial and the on-demand sub-trial (during 90 months).
Time Frame: After 90 months
Population: Safety Analysis Set includes all dosed subjects with data after dosing.
Measure: Number; unit: Number of Events
Arm/Group | Small Children (0 - <6 Years) | Older Children (6 - <12 Years) | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Number analyzed (Participants) | 27 | 28 | 23 | 135
Number of Events
  Adverse events | 180 | 204 | 240 | 636
  Serious adverse events | 6 | 8 | 6 | 27

3. Secondary Outcome: Annualised Bleeding Rate Reported During the Prevention Period (Only Applicable for Subjects in the Preventive Regimen)
Description: The number of bleeding episodes per year reported during the prevention period (during 90 months).
Time Frame: After 90 months
Population: Full Analysis Set. Number of subjects analysed=Subjects who received preventive regimen and were evaluable for the outcome.
Measure: Median (Full Range); unit: Bleeding episodes/year
Groups:
- Small Children (0 - <6 Years)-Preventive Regimen [Main Trial]: Subjects (0-<6 years) in main trial received turoctocog alfa (Preventive regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back to main trial before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or trial site was terminated by Novo Nordisk or relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009-30 Jun 2016). Preventive regimen: turoctocog alfa as slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly.
- Older Children (6 - <12 Years)-Preventive Regimen [Main Trial]: Subjects (6-<12 years) in main trial received turoctocog alfa (Preventive regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back to main trial before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg three times weekly or 40-60 IU/kg once every third day or twice weekly.
- Adolescents (12 - <18 Years)-Preventive Regimen [Main Trial]: Subjects (12-<18 years) in main trial received turoctocog alfa (Preventive regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back to main trial before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg three times weekly or 40-60 IU/kg once every third day or twice weekly.
- Adults (≥18 Years)-Preventive Regimen [Main Trial]: Subjects (>=18 years) in main trial received turoctocog alfa (Preventive regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back to main trial before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). Preventive regimen: Turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg three times weekly or 40-60 IU/kg once every third day or twice weekly.
Arm/Group | Small Children (0 - <6 Years)-Preventive Regimen [Main Trial] | Older Children (6 - <12 Years)-Preventive Regimen [Main Trial] | Adolescents (12 - <18 Years)-Preventive Regimen [Main Trial] | Adults (≥18 Years)-Preventive Regimen [Main Trial]
Number analyzed (Participants) | 27 | 28 | 23 | 129
Bleeding episodes/year | 1.08 [0 to 12.12] | 1.57 [0 to 10.8] | 1.57 [0 to 6.01] | 1.37 [0 to 17.82]

4. Secondary Outcome: Haemostatic Response to Turoctocog Alfa (None, Moderate, Good or Excellent) in Treatment of Bleeds.
Description: Haemostatic response to turoctocog alfa (none, moderate, good or excellent) in treatment of bleeds using a four-point response scale: none, moderate, good or excellent. The evaluation was done by patient, caregiver and/or investigator based on experience as follows: 1. Excellent: Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single infusion 2. Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after an infusion, but possibly requiring more than 1 infusion for complete resolution. 3. Moderate: Probable or slight beneficial effect within approximately 8 hours after the first infusion; usually requiring more than 1 infusion. 4. None: No improvement, or worsening of symptoms. This endpoint is measured during the preventive and on-demand sub-trial (during 90 months).
Time Frame: After 90 months
Population: Full Aanalysis Set. The endpoint was measured for preventive and on-demand regimen for comparison of the efficacy of turoctocog alfa between regimens. Number of subjects analysed=subjects who received preventive and on-demand regimen and were evaluable for this outcome.
Measure: Number; unit: Number of bleeds
Groups:
- Adolescents (12 - <18 Years) - Preventive Regimen [Main Trial]: Subjects (12-<18 years) in main trial received turoctocog alfa (Preventive regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back to main trial before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg three times weekly or 40-60 IU/kg once every third day or twice weekly.
- Adults (>= 18 Years) - Preventive Regimen [Main Trial]: Subjects (>=18 years) in main trial received turoctocog alfa (Preventive regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back to main trial before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). Preventive regimen: Turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day, 20-60 IU/kg three times weekly or 40-60 IU/kg once every third day or twice weekly.
- Adolescents (12-<18 Years)-(On-Demand Regimen [Main Trial]): Subjects (12-<18 Years) in main trial received turoctocog alfa (on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009-30 Jun 2016). On-Demand regimen: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment.
- Adults (>=18 Years)-(On-Demand Regimen [Main Trial]): Subjects (≥18 Years) in main trial received turoctocog alfa (on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). On-Demand regimen: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment.
- Adults (>=18 Years)-(On-Demand Regimen [Sub-trial]): Subjects (≥18 Years) in sub-trial received turoctocog alfa (on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. However during on-demand sub-trial, it was not possible for new subjects to switch to another regimen, subjects who did not comply with on-demand treatment regimen were to be withdrawn. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. Maximum treatment duration (27 Oct 2009 - 30 Jun 2016). On-Demand regimen: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment.
Arm/Group | Small Children (0 - <6 Years)-Preventive Regimen [Main Trial] | Older Children (6 - <12 Years)-Preventive Regimen [Main Trial] | Adolescents (12 - <18 Years) - Preventive Regimen [Main Trial] | Adults (>= 18 Years) - Preventive Regimen [Main Trial] | Adolescents (12-<18 Years)-(On-Demand Regimen [Main Trial]) | Adults (>=18 Years)-(On-Demand Regimen [Main Trial]) | Adults (>=18 Years)-(On-Demand Regimen [Sub-trial])
Number analyzed (Participants) | 21 | 24 | 22 | 103 | 1 | 7 | 14
Number of bleeds
  Excellent | 124 | 189 | 72 | 565 | 1 | 150 | 94
  Good | 62 | 103 | 103 | 382 | 6 | 22 | 105
  Moderate | 17 | 37 | 19 | 91 | 0 | 2 | 11
  None | 1 | 1 | 0 | 7 | 0 | 0 | 0
  Not known | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Missing | 0 | 1 | 2 | 5 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening (visit 1) starting after first exposure to Turoctocog alfa and until post treatment follow-up period (up to 90 months)
Description: The safety analysis set included all subjects exposed to turoctocog alfa
Groups:
- Small Children (0 - <6 Years): Subjects (0-<6 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day,20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
- Adolescents (12 - <18 Years): Subjects (12-<18 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day,20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
- Adults (≥18 Years): Subjects (≥18 years) received turoctocog alfa (preventive or on-demand regimen). Subjects switched between regimens during trial (main and on-demand sub-trial) upon investigators' discretion. Subjects coming from main trial were allowed to switch back before completion of 6 months on-demand regimen. Preventive regimen: turoctocog alfa as a slow iv bolus injection 20-50 IU/kg once every second day,20-60 IU/kg 3 times weekly or 40-60 IU/kg once every third day or twice weekly. On-Demand: Dose level aimed at a post injection level of at least 0.50 IU/mL of turoctocog alfa for treatment of bleeds as they occurred and occasionally as preventive treatment. All subjects were offered participation until either turoctocog alfa was commercially available in relevant country or until the trial, part of trial or a trial site was terminated by Novo Nordisk or a relevant authority for any reason in relevant country. The maximum treatment duration (27 Oct 2009 - 30 Jun 2016).
Arm/Group | Small Children (0 - <6 Years) | Older Children (6 - <12 Years) | Adolescents (12 - <18 Years) | Adults (≥18 Years)
Serious Adverse Events (participants affected / at risk) | 5/27 | 9/28 | 6/23 | 21/135
Other Adverse Events (participants affected / at risk) | 23/27 | 25/28 | 20/23 | 94/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Children (0 - <6 Years) (N=27) | Older Children (6 - <12 Years) (N=28) | Adolescents (12 - <18 Years) (N=23) | Adults (≥18 Years) (N=135)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device loosening (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal aneurysm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Children (0 - <6 Years) (N=27) | Older Children (6 - <12 Years) (N=28) | Adolescents (12 - <18 Years) (N=23) | Adults (≥18 Years) (N=135)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 1 (1) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 4 (7) | 19 (29)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 12 (13)
Bronchitis (Infections and infestations) | 1 (3) | 2 (2) | 2 (2) | 3 (3)
Chills (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 5 (8) | 4 (5) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 1 (1) | 4 (5) | 9 (11)
Dental caries (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (6) | 4 (19) | 5 (8) | 7 (8)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 3 (8) | 6 (29) | 17 (46)
Influenza (Infections and infestations) | 0 (0) | 2 (5) | 9 (13) | 9 (9)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (3) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (2) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 5 (19) | 1 (1) | 4 (5)
Limb injury (Injury, poisoning and procedural complications) | 1 (3) | 2 (3) | 4 (4) | 3 (4)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (4) | 5 (18) | 23 (41)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 14 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (2) | 7 (24) | 3 (9) | 9 (15)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 2 (6) | 5 (6) | 5 (6)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 2 (4) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (3) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (2)
Sinusitis (Infections and infestations) | 5 (6) | 1 (1) | 4 (7) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Tonsillitis (Infections and infestations) | 4 (8) | 2 (2) | 2 (6) | 2 (7)
Tooth development disorder (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 11 (12)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (9) | 5 (16) | 2 (2) | 16 (26)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (4) | 6 (6)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.